CLINICAL TRIAL: NCT01652183
Title: THE EFFECT OF INTRAOPERATIVE PARACETAMOL ON CATHETER-RELATED BLADDER DISCOMFORT: A PROSPECTIVE, RANDOMISED, DOUBLE-BLIND STUDY
Brief Title: Paracetamol for Catheter Related Bladder Discomfort
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pinar Ergenoglu (Other)
Responsible Party: Sponsor-Investigator, Pinar Ergenoglu, Baskent University School of Medicine Adana Teaching and Research Hospital, Baskent University
Organization: Baskent University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KA08/180
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Catheter Related Bladder Discomfort
Keywords: Intravenous paracetamol; catheter related bladder discomfort; urologic surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Control (n=32):iv 1.5 ml/kg 0.9% NaCl (Placebo Comparator)
  Interventions: Drug: Placebo
- Group Paracetamol(n=32):iv 15mg/kg paracetamol (Active Comparator): The patients were randomly divided into two groups: Group P (Paracetamol group, n=32) received intravenous 15mg/kg paracetamol during the surgery and Group C (Control Group, n=32) received intravenous 1.5 ml/kg 0.9% NaCl solution 30 minutes before the of surgery.At the end of the surgery, all patients had an nephrostomy catheter and the insertion site was infiltrated with 20 ml 0.25% bupivacaine infiltration for postoperative analgesia. Each patient received patient-controlled intravenous analgesia by meperidine (10 mg bolus, 20-minute lock-out, no infusion dose and 4 hour limit) for postoperative analgesia. All patients were planned to receive tenoxicam 20 mg intravenously as a rescue analgesic when visual analogue scale (VAS) was >3.
  Interventions: Drug: intravenous paracetamol

INTERVENTIONS:
Drug: intravenous paracetamol
  Other Names: 30.11.2005-118/79
  Arms: Group Paracetamol(n=32):iv 15mg/kg paracetamol
Drug: Placebo
  Arms: Group Control (n=32):iv 1.5 ml/kg 0.9% NaCl

SUMMARY:
The insertion of an urinary catheter in a patient undergoing a surgical procedure, especially in urinary interventions, may lead to catheter-related bladder discomfort with varying degrees of severity during the postoperative period. Catheter-related bladder discomfort (CRBD) symptoms associated with indwelling urinary catheter are similar to overactive bladder symptoms such as discomfort in the suprapubic region, urinary urgency, frequency, burning sensation with or without urge incontinence. Paracetamol is a drug with proven efficiency for the management of mild and moderate postoperative pain. In this study, the investigators hypothesized to address the effect of single-dose intravenous paracetamol on postoperative CRBD following percutaneous nephrolithotomy surgery (PNL).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age,
* American Society of Anesthesiologists (ASA) Physical Status of I-II,
* undergoing PNL with urinary bladder catheter.

Exclusion Criteria:

* obesity (BMI > 30),
* chronic opioid use,
* bladder outflow obstruction,
* benign prostatic hyperplasia, and
* overactive bladder (OAB) (frequency > 3 times at night or > 8 times within 24h).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Reducing of Catheter related bladder discomfort symptoms | CRBD was evaluated at postoperatively 30th minutes, 1st, 2nd, 4th, 6th and 12th hours
  CRBD was evaluated with a 4 point scale (1; no discomfort, 2; mild, revealed on questioning only, 3; moderate, stated by the patient without questioning, 4; severe, urinary urgency executed by behavioral responses, such as attempts to remove urinary catheter, restless extremity movements, verbal responses) at postoperatively 30th minutes, 1st, 2nd, 4th, 6th and 12th hours.

SECONDARY OUTCOMES:
Assessment of CRBD symptoms by the evaluation of VAS, sedation scales and hemodynamic findings | at postoperatively 30th minutes, 1st, 2nd, 4th, 6th and 12th hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University School of Medicine Adana Teaching and Research Hospital, Adana, Turkey (Türkiye)

REFERENCES:
- [Background] Agarwal A, Yadav G, Gupta D, Singh PK, Singh U. Evaluation of intra-operative tramadol for prevention of catheter-related bladder discomfort: a prospective, randomized, double-blind study. Br J Anaesth. 2008 Oct;101(4):506-10. doi: 10.1093/bja/aen217. Epub 2008 Jul 24. PMID 18653496
- [Background] Binhas M, Motamed C, Hawajri N, Yiou R, Marty J. Predictors of catheter-related bladder discomfort in the post-anaesthesia care unit. Ann Fr Anesth Reanim. 2011 Feb;30(2):122-5. doi: 10.1016/j.annfar.2010.12.009. Epub 2011 Jan 31. PMID 21277735
- [Derived] Ergenoglu P, Akin S, Yalcin Cok O, Eker E, Kuzgunbay B, Turunc T, Aribogan A. Effect of intraoperative paracetamol on catheter-related bladder discomfort: a prospective, randomized, double-blind study. Curr Ther Res Clin Exp. 2012 Dec;73(6):186-94. doi: 10.1016/j.curtheres.2012.08.001. PMID 24653520